CLINICAL TRIAL: NCT06468423
Title: Comparison of Deferasirox and Desferoxamine in Patients of β-Thalassemia Major With Iron Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESnTEC
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pateints of β-thalassemia Major With Iron Overload
MeSH Terms: interventions — Deferasirox; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deferasirox (DFX) group (Experimental): DFX group (n=71) included children who used oral (tablet) DFX at a dose of 30 mg/kg once daily for a duration of 6 months.
  Interventions: Drug: Deferasirox (DFX)
- Desferioxamine (DFO) group (Experimental): DFO group (n=71) included children who were given DFO at a dose of 50 mg/kg through the subcutaneous route by infusion pump five days a week
  Interventions: Drug: Deferoxamine (DFO)

INTERVENTIONS:
Drug: Deferasirox (DFX) — Oral DFX at a dose of 30mg/kg daily advised for a duration of 6 months.
  Other Names: Deferasirox
  Arms: Deferasirox (DFX) group
Drug: Deferoxamine (DFO) — DFO group (n=71) included children who were given DFO at a dose of 50 mg/kg through the subcutaneous route by infusion pump five days a week for a duration of 6 months.
  Other Names: Deferoxamine
  Arms: Desferioxamine (DFO) group

SUMMARY:
This study was planned to compare deferasirox and desferrioxamine in terms of mean serum ferritin levels in patients of β-thalassemia major having Iron overload. Choosing an effective iron chelator is crucial to increasing iron chelation therapy compliance. Not much local data exists in Pakistan comparing the effectiveness of deferasirox (DFX) and desferrioxamine (DFO), so, this study would be helpful in providing baseline data and formulating new protocols for iron chelation therapy, in which DFX may be a useful oral alternative to parenteral DFO.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of β-thalassemia major (as per medical record or confirmed by hemoglobin electrophoresis)
* Iron overload (serum ferritin level above 1000 µg/L)

Exclusion Criteria:

* Patients with other transfusion-dependent anemias
* Thalassemia major with cardiomyopathy or arrhythmia.
* Chronic renal failure
* Chronic liver disease (ALT >200 IU)
* Hhypersensitivity to deferasirox or desferrioxamine
* Patients already on combined chelation therapy

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Mean Serum Ferritin Levels | 6 months
  Change in mean serum ferritin level from baseline for each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Thalassemia Center of Hematology Department, The Children's Hospital & The Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable resquest to parimary researcher.